CLINICAL TRIAL: NCT03652766
Title: A Pilot and Feasibility Study of Daily Weight Tracking to Manage Gestational Weight Gain During Pregnancy
Brief Title: Pregnancy Weight Tracking Pilot Project
Acronym: PTRK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FWA00000312-9
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Obesity Complicating Childbirth
Keywords: Overweight; Obesity; e-Health; Gestational Weight Gain; Pregnancy; Women's Health; Prevention
MeSH Terms: conditions — Overweight; Obesity; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Single group feasibility and acceptability trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily Weight Tracking (Other): Participants will be provided with a wireless Bluetooth-enabled bathroom scale with instructions for connecting it to their home wifi network or phone using Bluetooth and a mobile app, and will also be walked through creating an anonymous study account for app access. They will be asked to track their weight daily for 6 weeks and will receive weekly feedback on weight gain trajectories along with nutrition or physical activity messages for healthy pregnancy weight gain.
  Interventions: Behavioral: Daily Weight Tracking

INTERVENTIONS:
Behavioral: Daily Weight Tracking — Daily weight tracking + weekly email or text message feedback

SUMMARY:
This pilot study will examine perceptions about daily weighing for pregnant women with overweight or obesity by testing the feasibility, acceptability, and preliminary efficacy of daily weighing for reducing excess gestational weight gain (GWG) within the context of a low intensity, digital-health based intervention delivered remotely with electronic feedback to participants.

DETAILED DESCRIPTION:
Excessive weight gain during pregnancy is predictive of a host of health outcomes in both the mother and child, particularly among women who are overweight or obese pre-pregnancy. Gaining too much weight is associated with higher risk of gestational diabetes, large birth weight for the baby and its corresponding risks, and postpartum obesity. Alarmingly, these outcomes persist for years after birth. For adults who are overweight or obese and interested in weight management, a key element of behavioral weight control is self-monitoring. Supported by self-regulation theory, the effectiveness of daily weighing is likely a function of the self-regulatory processes that are activated as a result of this behavior. Receiving feedback daily on weight proximal to diet and exercise behaviors may increase awareness how of behaviors impact weight and allow for small changes in weight to be understood and resolved through subsequent behavior change. Given the improvements in self-regulation as a result of daily weighing, it may be an effective strategy for reducing excessive gestational weight gain during pregnancy. It is not clear, however, whether pregnant women would engage in this behavior and whether daily weighing would be effective in promoting recommended levels of weight gain during pregnancy.

To determine the feasibility of a six-week, digital health daily weighing pilot intervention to monitor gestational weight gain among overweight and obese pregnant women, participants will be recruited at up to 20 weeks' gestation (consistent with prior studies) and will receive a digital wireless Bluetooth-enabled scale to track weight for six weeks during pregnancy. They will receive tailored feedback via weekly emails in response to adherence to daily weighing and whether weight gains are in accordance with recommended levels and healthy standards for pregnancy; weekly emails will also communicate healthy eating and physical activity tips for pregnancy. They will be asked to complete surveys at baseline (before using scales) and follow-up (after using scales) that focus on experiences with weight monitoring, GWG knowledge and expectations, and perceptions of the intervention process.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35
* Up to 20 weeks' gestation in their first pregnancy
* Low-risk uncomplicated pregnancy
* Have overweight or obesity just prior to becoming pregnant
* Have an iPhone or Android smartphone with wireless/Bluetooth capability

Exclusion Criteria:

* Individuals who are not pregnant
* Second or subsequent pregnancy
* No iPhone or Android smartphone with Bluetooth capacity
* No wifi network at home
* Expecting twins or other multiple
* More than 20 weeks gestation
* High-risk or complicated pregnancy for which participation would be contraindicated
* Of advanced maternal age according to obstetric guidelines (i.e., age 36 or older)
* Diabetes or history of eating disorders
* Pre-pregnancy weight less than 25 kg/m2 or greater than 36 kg/m2 (either not overweight or with extreme obesity)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Adherence (protocol feasibility) | 6 weeks
  Frequency of bathroom scale use under daily weight tracking instruction condition

SECONDARY OUTCOMES:
Acceptability (protocol) | 6 weeks
  Preferences and beliefs regarding daily weight tracking instruction condition
Gestational Weight Gain | 6 weeks
  Weight gain during pregnancy under daily weight tracking instruction condition
Gestational Weight Gain Knowledge | 6 weeks
  Use of bathroom scale and understanding of recommendations for gestational weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Linde, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to the link between identifiers (name and date of birth) and participants study ID numbers, which will be kept on paper in a locked file cabinet in a private office, will be limited to the investigator; only de-identified datasets will be shared with future grant submission collaborators as needed, and those files will be password-protected and shared via encrypted transmission.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be shared until the related NIH grant is submitted, for a period of no longer than one year.
Access Criteria: Collaborators on NIH grant proposal submission for 2019.